CLINICAL TRIAL: NCT00526916
Title: PET Imaging of Peripheral Benzodiazepine Receptors in Patients With Neurocysticercosis Using [C-11]PBR28
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 070208; 07-M-0208
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-09-05

CONDITIONS: Neurocysticercosis; Healthy
Keywords: Epilepsy; Taenia Solium; Microglia; Neuroinflammation; Compartment Model; Neurocysticercosis; Healthy Volunteer; HV
MeSH Terms: conditions — Neurocysticercosis; Epilepsy; Taeniasis; Neuroinflammatory Diseases

INTERVENTIONS:
Drug: [C-11]PBR28

SUMMARY:
The purpose of this protocol is to measure peripheral benzodiazepine receptors in the brain using positron emission tomography (PET) and compare the imaging results between patients and healthy people.

DETAILED DESCRIPTION:
Objective

In endemic regions neurocysticercosis is the most common cause of adult acquired epilepsy and thus an important public health problem. The disease is caused by infection with the larval form of the tapeworm, Taenia solium. Although neurocysticercosis is common only in many developing regions, an increased number of patients are diagnosed in developed countries mostly due to immigration of infected individuals.

The peripheral benzodiazepine receptor (PBR) can be a clinically useful marker to detect neuroinflammation because activated microglia in inflammatory areas expresses much greater levels of PBR than in microglia in resting conditions. PBR has been imaged with positron emission tomography (PET) using [(11)C]1-(2-chlorophenyl-N-methylpropyl)-3-isoquinoline carboxamide (PK11195), which provides low levels of specific signal. Recently we developed a new ligand, [(11)C]N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine (PBR28), which showed much greater specific signal than [(11)C]PK11195 in non-human primates.

The major objective of this protocol is to assess the utility of [(11)C]PBR28 PET to detect neuroinflammation in patients with neurocysticercosis.

Study population

Thirty patients will be recruited and clinically followed under protocol 85-I-0127, Treatment of Cysticercosis including Neurocysticercosis with Praziquantel or Albendazole, (PI: Theodore E. Nash, MD, NIAID). Thirty healthy subjects will be recruited.

Design

Fifteen patients with neurocysticercosis and the first 15 age-matched healthy subjects will have brain PET scans. Patients will have up to three [(11)C]PBR28 PET scans during the follow-up and the treatment under 85-I-0127, typically a few weeks apart.

Outcome measures

PBR28 binding will be compared with clinical symptoms and MRI findings. In addition, the binding will be compared between patients and age-matched control subjects because the high levels of specific binding may allow detection of an increase of PBR in regions where MRI does not detect inflammation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Common to patients with neurocysticercosis and healthy subjects:

Ages between 18 and 75, inclusive.

Patients must meet the inclusion criteria of protocol 85-I-0127.

CONTROL SUBJECTS:

Are healthy based on history, physical exams, ECG, and lab tests.

EXCLUSION CRITERIA:

COMMON TO ALL SUBJECTS:

Current psychiatric illness, substance abuse or severe systemic disease based on history and physical exam.

ECG with clinically significant abnormalities. Any existing physical exam and ECG within one year will be reviewed and if none already exists in the chart, these will be obtained and reviewed.

Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual guideline of RSC.

Pregnancy or breast feeding.

Claustrophobia.

Positive HIV test.

Cannot lie on back for a few hours for the PET scans.

Presence of ferromagnetic metal in the body or heart pacemaker.

ADDITIONAL EXCLUSION CRITERIA FOR PATIENTS:

Medically unstable.

Seizures are not well controlled with medications.

A history of brain disease other than neurocysticercosis.

Laboratory tests with clinically significant abnormalities unrelated to neurocysticercosis or its treatment.

ADDITIONAL EXCLUSION CRITERIA FOR HEALTHY SUBJECTS:

Laboratory tests with clinically significant abnormalities.

A history of brain disease.

The usage of nonsteroidal and other anti-inflammatory medications is not an exclusion criterion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-09-04; Study Completion 2014-09-05 (Actual)

PRIMARY OUTCOMES:
Binding of [C-11]PBR28 at peripheral benzodiazepine receptors

SECONDARY OUTCOMES:
MRI | years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Anholt RR, Murphy KM, Mack GE, Snyder SH. Peripheral-type benzodiazepine receptors in the central nervous system: localization to olfactory nerves. J Neurosci. 1984 Feb;4(2):593-603. doi: 10.1523/JNEUROSCI.04-02-00593.1984. PMID 6321699
- [Background] Anholt RR, Pedersen PL, De Souza EB, Snyder SH. The peripheral-type benzodiazepine receptor. Localization to the mitochondrial outer membrane. J Biol Chem. 1986 Jan 15;261(2):576-83. PMID 3001071
- [Derived] Paul S, Gallagher E, Liow JS, Mabins S, Henry K, Zoghbi SS, Gunn RN, Kreisl WC, Richards EM, Zanotti-Fregonara P, Morse CL, Hong J, Kowalski A, Pike VW, Innis RB, Fujita M. Building a database for brain 18 kDa translocator protein imaged using [11C]PBR28 in healthy subjects. J Cereb Blood Flow Metab. 2019 Jun;39(6):1138-1147. doi: 10.1177/0271678X18771250. Epub 2018 May 11. PMID 29749279